CLINICAL TRIAL: NCT05220085
Title: Real-life Beovu Experience at UZ Leuven for the Treatment of Exudative Neovascular Age-related Macular Degeneration
Brief Title: Beovu Experience UZ Leuven
Acronym: BEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, JulieJacob, prof.dr.Julie Jacob, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S66240
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Brolucizumab Ophthalmic Dbll 6 Mg/0.05 mL Intravitreal Solution — Intravitreal injection

SUMMARY:
Reporting early real-world clinical data of consecutive patients on the use of Beovu® (brolucizumab) intravitreal injections in patients with neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
Brolucizumab (Beovu, Novartis, Basel, Switzerland) is the newest anti-vascular endothelial growth factor (anti-VEGF) drug. It received FDA approval for the treatment of neovascular age-related macular degeneration (nAMD) in October 2019 followed by EMA approval in February 2020. Brolucizumab received marketing approval based on the two pivotal phase 3 clinical trials - HAWK and HARRIER - with a q8/q12 week dosing regimen. Potential benefits of brolucizumab are assumed to be related to its low molecular weight with subsequent better tissue penetration as well as higher molar concentration. This could improve the treatment durability and lower the burden for patients and caregivers when dealing with repetitive intravitreal treatments and monitoring visits over a long period of time in a chronic disease. However, safety signals have been reported in both RCTs and post-marketing reports, which included the occurrence of intraocular inflammation (IOI) and retinal vasculitis with or without occlusion.

In this study we want to share our early results and experience with Bolucizumab in UZ Leuven. By retrospective analysis of a cohort of 17 patients treated with Brolucizumab, we evaluate the efficacy of the drug as well as the occurrence of adverse-events, especially intra-ocular inflammation and vasculitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of neovascular age-related macular degeneration
2. Partial response on current anti-VEGF treatment or unability to prolong the treatment interval beyond 6 or 8 weeks

Exclusion Criteria:

* 1. Any form of previous intraocular inflammation 2. Any form of previous inflammatory reaction after anti-VEGF treatment 3. Functionally monophthalmic patients 4. Any sign of active intraocular inflammation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants eligible for inclusion in this Study must meet all of the following criteria:
  1. Diagnosis of neovascular age-related macular degeneration
  2. Partial response on current anti-VEGF treatment or unability to prolong the treatment interval beyond 6 or 8 weeks
  List details under which a participant is considered unsuitable for inclusion in the Study.
  Participants eligible for this Study must not meet any of the following criteria:
  1. Any form of previous intraocular inflammation
  2. Any form of previous inflammatory reaction after anti-VEGF treatment
  3. Functionally monophthalmic patients
  4. Any sign of active intraocular inflammation
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
anatomical efficacy of treatment with brolucizumab | dec 2020- nov 2021
  central retinal thickness
functional efficacy of treatment with brolucizumab | dec 2020- nov 2021
  best corrected visual acuity

SECONDARY OUTCOMES:
Safety of treatment with brolucizumab | dec 2020- nov 2021
  Safety: occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Julie Jacob, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLEUVEN, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dugel PU, Koh A, Ogura Y, Jaffe GJ, Schmidt-Erfurth U, Brown DM, Gomes AV, Warburton J, Weichselberger A, Holz FG; HAWK and HARRIER Study Investigators. HAWK and HARRIER: Phase 3, Multicenter, Randomized, Double-Masked Trials of Brolucizumab for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Jan;127(1):72-84. doi: 10.1016/j.ophtha.2019.04.017. Epub 2019 Apr 12. PMID 30986442
- [Background] Dugel PU, Singh RP, Koh A, Ogura Y, Weissgerber G, Gedif K, Jaffe GJ, Tadayoni R, Schmidt-Erfurth U, Holz FG. HAWK and HARRIER: Ninety-Six-Week Outcomes from the Phase 3 Trials of Brolucizumab for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2021 Jan;128(1):89-99. doi: 10.1016/j.ophtha.2020.06.028. Epub 2020 Jun 20. PMID 32574761
- [Background] Dugel PU, Jaffe GJ, Sallstig P, Warburton J, Weichselberger A, Wieland M, Singerman L. Brolucizumab Versus Aflibercept in Participants with Neovascular Age-Related Macular Degeneration: A Randomized Trial. Ophthalmology. 2017 Sep;124(9):1296-1304. doi: 10.1016/j.ophtha.2017.03.057. Epub 2017 May 24. PMID 28551167
- [Background] Holz FG, Dugel PU, Weissgerber G, Hamilton R, Silva R, Bandello F, Larsen M, Weichselberger A, Wenzel A, Schmidt A, Escher D, Sararols L, Souied E. Single-Chain Antibody Fragment VEGF Inhibitor RTH258 for Neovascular Age-Related Macular Degeneration: A Randomized Controlled Study. Ophthalmology. 2016 May;123(5):1080-9. doi: 10.1016/j.ophtha.2015.12.030. Epub 2016 Feb 20. PMID 26906165
- [Background] Witkin AJ, Hahn P, Murray TG, Arevalo JF, Blinder KJ, Choudhry N, Emerson GG, Goldberg RA, Kim SJ, Pearlman J, Schneider EW, Tabandeh H, Wong RW. Occlusive Retinal Vasculitis Following Intravitreal Brolucizumab. J Vitreoretin Dis. 2020 Jul;4(4):269-279. doi: 10.1177/2474126420930863. Epub 2020 Jul 1. PMID 32789284
- [Background] Jain A, Chea S, Matsumiya W, Halim MS, Yasar C, Kuang G, Sepah YJ, Khanani AM, Do DV, Nguyen QD. Severe vision loss secondary to retinal arteriolar occlusions after multiple intravitreal brolucizumab administrations. Am J Ophthalmol Case Rep. 2020 Apr 2;18:100687. doi: 10.1016/j.ajoc.2020.100687. eCollection 2020 Jun. PMID 32280811
- [Background] Baumal CR, Spaide RF, Vajzovic L, Freund KB, Walter SD, John V, Rich R, Chaudhry N, Lakhanpal RR, Oellers PR, Leveque TK, Rutledge BK, Chittum M, Bacci T, Enriquez AB, Sund NJ, Subong ENP, Albini TA. Retinal Vasculitis and Intraocular Inflammation after Intravitreal Injection of Brolucizumab. Ophthalmology. 2020 Oct;127(10):1345-1359. doi: 10.1016/j.ophtha.2020.04.017. Epub 2020 Apr 25. PMID 32344075
- [Background] Haug SJ, Hien DL, Uludag G, Ngoc TTT, Lajevardi S, Halim MS, Sepah YJ, Do DV, Khanani AM. Retinal arterial occlusive vasculitis following intravitreal brolucizumab administration. Am J Ophthalmol Case Rep. 2020 Mar 31;18:100680. doi: 10.1016/j.ajoc.2020.100680. eCollection 2020 Jun. PMID 32258827
- [Background] Sharma A, Kumar N, Parachuri N, Singh S, Bandello F, Kuppermann BD, Loewenstein A. Brolucizumab-related retinal vasculitis: emerging disconnect between clinical trials and real world. Eye (Lond). 2021 May;35(5):1292-1294. doi: 10.1038/s41433-020-01227-w. Epub 2020 Oct 20. No abstract available. PMID 33082532
- [Background] Mones J, Srivastava SK, Jaffe GJ, Tadayoni R, Albini TA, Kaiser PK, Holz FG, Korobelnik JF, Kim IK, Pruente C, Murray TG, Heier JS. Risk of Inflammation, Retinal Vasculitis, and Retinal Occlusion-Related Events with Brolucizumab: Post Hoc Review of HAWK and HARRIER. Ophthalmology. 2021 Jul;128(7):1050-1059. doi: 10.1016/j.ophtha.2020.11.011. Epub 2020 Nov 15. PMID 33207259
- [Background] Holz FG, Heinz C, Wolf A, Hoerauf H, Pleyer U. [Intraocular inflammation with brolucizumab use : Patient management-diagnosis-therapy]. Ophthalmologe. 2021 Mar;118(3):248-256. doi: 10.1007/s00347-021-01321-8. Epub 2021 Feb 8. German. PMID 33555415